CLINICAL TRIAL: NCT06616363
Title: (PAG POTS - NIH) Pediatric Postural Orthostatic Tachycardia Syndrome (POTS) : Does a Periaqueductal Gray-vagus Nerve Interface Malfunction Explain the Natural History With Its Numerous Co-morbidities?
Brief Title: Does a Periaqueductal Gray-vagus Nerve Interface Malfunction Explain the Nat hx With Its Numerous Co-morbidities?
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20029682; 1R01HL163577 (NIH)
Record Dates: First submitted 2024-07-23; First posted 2024-09-27 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: POTS - Postural Orthostatic Tachycardia Syndrome
Keywords: PAG activation; Cardiovagal Modulation
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — -Stool samples will be sent for analysis, they will then be de-identified and stored in a -80 C freezer at VCU for future research purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 60 POTS Postural Tachycardia Syndrome (POTS): POTS patients will be current patients of the study practitioners within the autonomic, cardiology PM&R clinics and autonomic laboratory. This cohort may receive a codified treatment plan within the following 7 treatment categories which are also standard of care procedures based on clinical recommendations: (1) salt, fluid and diet management; (2) exercise program with or without PT; (3) cognitive behavioral therapy or other counseling; (4) vagal stimulation forms like yoga, breathing exercises, relaxation, microauricular stimulation; (5) pharmacotherapy for pressure maintenance; (6) medications for pain and headache; (7) medications for the gastrointestinal issues.
  Interventions: Behavioral: Questionnaires to be competed; Behavioral: Provide list of medication and lifetime events; Behavioral: Use phone App to record new life events; Device: Will wear an activity monitor; Other: Periodic 24-hour urine sodium check; Diagnostic Test: A fMRI scan; Diagnostic Test: A bedside tilt test will be performed; Other: IV placed to collect blood samples; Other: Stool Sample
- 40 Post-Infection cohort: Post-Infection participants will be identified through Best Practice Alerts through EPIC, and referrals from hospitalist and gastroenterology inpatient services. Post-Infection cohorts will be approached up to 6 weeks after they are released from the hospital, to ensure they are healthy enough to participate.
  Interventions: Behavioral: Questionnaires to be competed; Behavioral: Provide list of medication and lifetime events; Behavioral: Use phone App to record new life events; Device: Will wear an activity monitor; Diagnostic Test: A fMRI scan; Diagnostic Test: A bedside tilt test will be performed; Other: IV placed to collect blood samples; Other: Stool Sample
- 20 healthy controls: Healthy control participants will be recruited from local communities using flyers, social media and using EPIC Best Practice Alerts.
  Interventions: Behavioral: Questionnaires to be competed; Behavioral: Provide list of medication and lifetime events; Behavioral: Use phone App to record new life events; Device: Will wear an activity monitor; Diagnostic Test: A fMRI scan; Diagnostic Test: A bedside tilt test will be performed; Other: IV placed to collect blood samples; Other: Stool Sample

INTERVENTIONS:
Behavioral: Questionnaires to be competed — * The Pain Coping Questionnaire short form
  * Functional Disability Inventory (FDI), the primary clinical outcome measure.
  * COMPASS-31 and orthostatic hypotension modified for POTS.
  * The Pain Response Inventory (PRI)PROMIS Depression
  * GAD-7 for anxiety
  * Varni/Thompson Pediatric Pain Questionnaire
  * Child and Parent Reports of Post-Traumatic Symptoms (CROPS/PROPS)
  * Pain Catastrophizing Scale (PCS-C)
  * Detailed account of natural history and evolution of POTS and COPCs through MEDYSA (facilitates the assessment of specific syndromic diagnoses based on published criteria, rather than organ-based classification of symptoms)
Behavioral: Provide list of medication and lifetime events — Participants will provide a list of all medications taken at each visit time, lifetime history of infections, traumas, and other significant life events.
Behavioral: Use phone App to record new life events — Subjects will also record new life events, minor traumas, entrance into a flare and menses in Ilumivu's EMA (Ecological Momentary Assessment) phone App
Device: Will wear an activity monitor — Participants will have an activity monitor loaned for the duration of the study to track their physical activity.
Other: Periodic 24-hour urine sodium check — POTS patients will have a periodic 24-hour urine sodium check to determine compliance to intake of salt.
  Groups: 60 POTS Postural Tachycardia Syndrome (POTS)
Diagnostic Test: A fMRI scan — • Participants will complete a fMRI scan without contrast and complete a looming animacy threat task; participants judge the valence of images via button press as they perceive the image.
Diagnostic Test: A bedside tilt test will be performed — A bedside tilt test will be performed where blood pressure will be recorded supine and upright positions to confirm/exclude POTS.
Other: IV placed to collect blood samples — • An IV will be place for collection of 4 blood samples, about 12 mL of blood. For each position (lying and standing) the study team will draw 2 tubes each times with 3 mL of blood, for a total of 4 lab tubes (12 mL). Physical exams to assess the 18-tender points described by the American College of Rheumatology for the diagnosis of fibromyalgia and hypermobility/Ehlers-Danlos Syndrome (EDS) exam will be performed in all subjects.
Other: Stool Sample — • Participants will provide a stool biospecimen sample at each in-person visit. Stool will be collected in a hat and sample will be swabbed with the swab placed directly into PrimeStore collection tube and the remainder of the sample discarded

SUMMARY:
Postural tachycardia syndrome (POTS) is a common and disabling disorder among adolescents. No epidemiologic data exist to support the often cited 0.5 to 2% prevalence. Case series suggest 3 to 5 times greater incidence in girls than boys. POTS is defined in children as daily chronic symptoms of orthostatic intolerance and a 40 bpm rise in heart rate in the first 10 minutes of a tilt study in the absence of orthostatic hypotension. POTS often develops after an acute event like an illness, infection, immunization, head trauma, psychological trauma or surgery. Natural history data are absent for POTS, though some outcome studies exist. Orthostatic symptoms improve in the majority and heart rate changes improve in 38% at 1 year. A 2-year follow up showed small improvement in comorbid symptoms of POTS in a 12 subject cohort followed yearly. In a pediatric 5-year outcome follow up questionnaire study, 86% of adolescents with POTS reported resolved, improved, or intermittent, symptoms, with primarily physical rather than mental health complaints.

DETAILED DESCRIPTION:
The current definition of POTS highlights the peripheral mechanistic emphasis of 30 years of studies exploring cardio- and cerebro-vascular, immunologic, mast cell activation, connective tissue and other physiologic mechanisms. The classification of POTS itself also assumes a peripheral etiology, typically including neuropathic, hyperadrenergic, hypovolemic and sometimes immune POTS. However, a central nervous system (CNS) etiology might better account for what is knowns about POTS currently: (1) POTS often follows an infection, physical or psychological trauma. (2) POTS occurs most often in post-menarche adolescent girls volume redistribution differs across subjects (4) exercise, cognitive behavioral therapy provide best long-term outcomes (5) co-morbid disorders, typically overlapping pain conditions such as migraine headache, fibromyalgia, and most functional gastrointestinal disorders (FGID), often dominate the clinical picture. COPCs are typically considered to reflect a CNS etiology.

Because it coordinates the autonomic, motor and pain responses to an acute threat, the midbrain periaqueductal gray region (PAG) is an attractive candidate whose dysfunction could potentially explain all major features of POTS, including the frequent antecedent emotional or physical threat, the POTS core autonomic changes, and the co-morbid pain disorders. The PAG interprets threats as escapable or inescapable, specifically activating a different column for each response type.

ELIGIBILITY:
POTS sample

Inclusion Criteria:

* symptomatic ≥ 40 bpm rise in heart rate in the first 10 min of a tilt table study without a drop in blood pressure
* Clinical symptoms of orthostatic intolerance

Exclusion Criteria:

* Pregnant or breastfeeding
* Cognitive defects that preclude answering questionnaires or following assessment directions
* Other chronic diseases
* Unstable medical conditions
* Use of narcotics
* Limited English proficiency
* Investigator discretion that participant would not be suitable to participate
* A phone older than 5 years old or unable to support EMA software

POST INFECTION

Inclusion Criteria:

* acute upper respiratory or gastrointestinal infection that required admission to the acute care units but not requiring an ICU stay

Exclusion Criteria:

* Pregnant or breastfeeding
* Chronic prescriptions, history of POTS or orthostatic symptoms, recent inpatient psychiatric admissions, substance use disorder, trauma such as a motor vehicle accident, surgery, or other significant physical or emotional trauma in the last 5 years
* Cognitive defects that preclude answering questionnaires or following assessment directions
* Other unstable chronic diseases
* Unstable medical conditions
* Use of narcotics
* Severe depression or anxiety (untreated / unstable)
* Limited English proficiency
* Investigator discretion that participant would not be suitable to participate
* A phone older than 5 years old or unable to support EMA software

HEALTHY CONTROLS

Inclusion Criteria:

* Apparently healthy with no known chronic illnesses

Exclusion Criteria:

* Pregnant or breastfeeding
* History of POTS or orthostatic symptoms, migraines, fibromyalgia, chronic fatigue, PTSD. Functional gastrointestinal disorders, fainting, dysmenorrhea, or other chronic pain syndrome, inpatient psychiatric admissions, substance use disorder, trauma such as a motor vehicle accident, surgery, or other significant physical or emotional trauma in the last 5 years
* Cognitive defects that preclude answering questionnaires or following assessment directions
* Other chronic unstable diseases
* Unstable medical conditions
* Use of narcotics
* Severe depression or anxiety (untreated / unstable)
* Limited English proficiency
* Investigator discretion that participant would not be suitable to participate
* A phone older than 5 years old or unable to support EMA software

Ages: 12 Years to 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only females aged 12-21. Females will be targeted specifically since POTS is more common in females than males and avoids creation of a subgroup too small to analyze.
Study Population: The study aims to recruit only females aged 12-21. Females will be targeted specifically since POTS is more common in females than males and avoids creation of a subgroup too small to analyze.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-05-29 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Functional Disability Inventory (FDI) | Experimental Cohort: Baseline and monthly for 24 months (3, 6, 12, 24 in-person study visits), the other months will be completed from home. The control cohort: months 0-12
  The total score determines the level of functional disability, in which higher numbers represent a higher level of disability. There are 15-items and a score of 0 indicates that there are no complaints present whereas 30 indicates that the patient is extremely disabled. The Functional Disability Inventory (FDI) is one of the most widely used measures of functional impairment among children and adolescents with chronic pain. It is expected that there will be higher threat sensitivity that correlates with POTS severity (FDI score) across the POTS cohort, and within subjects based on clinical evolution.
Pain Coping Questionnaire short form | Experimental Cohort: Baseline and monthly for 24 months (3, 6, 12, 24 in-person study visits), the other months will be completed from home. The control cohort: months 0-12
  The Pain Coping Questionnaire (PCQ) is a 39-item self-report measure for evaluating pain coping in children and adolescents in both clinical and research settings. It consists of 8 subscales that can be categorized into 3 higher-order factors, including approach (composed of information seeking, problem-solving, and seeking social support subscales), problem-focused avoidance (composed of positive self-statements, behavioural distraction, and cognitive distraction subscales), and emotion-focused avoidance (composed of externalizing and internalizing/catastrophizing subscales). Higher scores indicate higher use of a particular coping strategy or style.
Pain Catastrophizing Scale (PCS-C) | Experimental Cohort: Baseline and monthly for 24 months (3, 6, 12, 24 in-person study visits), the other months will be completed from home. The control cohort: months 0-12
  The Pain Catastrophizing Scale for Children (PCS-C) is a 13-item self-report scale that measures how children think negatively about pain. The PCS-C asks respondents to rate how often they have pain-related thoughts and feelings on a scale of 0-4, with 0 meaning "not at all true" and 4 meaning "very true". The PCS-C is scored 1) Total score: The sum of all responses, ranging from 0-52, with higher scores indicating more catastrophic thinking 2) Subscale scores: The PCS-C assesses three dimensions of pain catastrophizing: rumination, magnification, and helplessness
Functional MRI (fMRI) scan while completing a complete a looming animacy threat task; participants judge the valence of images via button press as they perceive the image. | Experimental cohort: Baseline, 3, 6, 12, 24 month in person visits. Control Cohort: Baseline, 3, 6, and 12 month in person visits.
  Functional MRI is a type of MRI scan that can show which areas of your brain are most active. Tracking and comparing that activity to what you were doing at the time can help "map" your brain activity. It's most often used for planning surgery or similar procedures in the brain. Functional MRI (fMRI) scan in this study will be completed while completing a looming animacy threat task; participants judge the valence of images via button press as they perceive the image.
Bedside Tilt test | Experimental cohort: Baseline, 3, 6, 12, 24 month in person visits. Control Cohort: Baseline, 3, 6, and 12 month in person visits.
  A tilt table test, also known as a tilt test, is a procedure that helps determine the cause of fainting or near fainting spells. It involves lying on a table that's tilted to different positions while a medical professional monitors your heart rate, blood pressure, and oxygen levels.

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Chelimsky, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States